CLINICAL TRIAL: NCT01899443
Title: Improving Services and Outcomes for Joint Replacement Patients
Status: Completed | Type: Observational
Sponsor: South West Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Justine Naylor, Senior Principal Research Fellow; Director, South West Sydney Local Health District
Other Study IDs: ISOAJRS_AU
Record Dates: First submitted 2013-07-10; First posted 2013-07-15 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis
Keywords: total hip replacement; total knee replacement; patient outcomes; health services research
MeSH Terms: conditions — Osteoarthritis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total hip and knee replacement patients: This study will select up to 20 high volume (>275 cases annually) public and private hospitals across Australia. A random sample of c.2200 patients with diagnosis of osteoarthritis undergoing primary total hip or knee replacement surgery will be recruited.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — This is an observational study observing relationship between routine care and outcomes after total hip or knee arthroplasty.

SUMMARY:
Primary total knee or total hip replacement surgeries are costly high volume procedures & outcomes may be affected by surgical & care processes & individual patient characteristics. The primary hypotheses is that non compliance with recommended practice impacts patient outcomes (e.g. the likelihood of complications following surgery). The primary aims of the study are to evaluate the links between processes & outcomes & if possible develop a model that will improve patient outcomes & reduce unnecessary practice variation whilst considering costs.

DETAILED DESCRIPTION:
The primary aim of the study is to identify whether compliance with specific processes is associated with better outcomes.

The study is a longitudinal cohort study to examine outcomes after total hip and knee replacement surgeries. We hypothesise the site and patient level compliance is related to the prevalence of a subsequent complication (composite outcome comprising 30 day mortality, readmission, reoperation or surgical complication).

METHODS This study will select high volume (>275 cases annually) public and private hospitals across Australia. By involving public and private sites across Australia, the generalisability of the findings is enhanced. Each site will identify a site coordinator to oversee and manage the project at that site. Site coordinators are identified by each site. After hospital discharge, patients are followed up by the investigators.

This is a prospective observational study with projected sample of c.2200 consenting patients from up to 20 high volume hospitals. The site coordinator will screen, approach and consent eligible patients during routine preadmission processes. At the time of consent, the patient will be required to: provide socio-demographic details about themselves, past medical history, complete 2 standard patient reported outcome measures. Contact with patients about the study will be made by the site coordinator and routine hospital staff involved in their acute care. Acute data collection will involve prospective audit of medical records to collect peri- and post- operative acute care process data, client characteristics and outcomes by staff at each site. Random and convenience sampling will be used to identify eligible hospital sites which will remain anonymous.

Patient follow up regarding longer term outcomes will be completed via telephone by study investigators at three additional time points (approximately 35 and 90 days and 1 year post surgery) to collect repeat data as provided by each patient at the time of consent.

Descriptive statistics will be used to profile site level and patient level compliance with key processes of care. Multivariable logistic regression (MLoR) will be used to identify the association between the binary composite outcome measure and patient level compliance. Site and individual patient compliance with evidence based guidelines (where available) or best practice recommendations on key processes and relevant outcomes will be examined (e.g. Venous thromboembolism (VTE) prevention). Sample size calculations have been completed to ensure the analyses have sufficient power. If a useful association between processes and outcomes is identified, cost analyses with specific foci will be undertaken to consider costs for different factors and stages (e.g. acute / post discharge). Secondary analysis will determine the predictors of patient -reported outcomes. Depending on the results of initial data analyses, additional secondary analyses will potentially include analyses at additional time points (beyond initial 35 days) for association between key processes and outcomes, and analysis looking at the association between specific complications and compliance with specific processes.

Interim analysis will be undertaken to assess the level of observed compliance with key processes.

Re-abstraction of acute care data will be undertaken to ensure accuracy and completeness of submitted date from the sites.

Site survey Prior to study commencement at each site, the site coordinators will complete a survey detailing each surgeons protocols for key processes including their VTE and antimicrobial prophylaxes. The extent surgeon protocols align with Australian practice guidelines will be ascertained.

Additional secondary analyses will include, but may not be limited to:

1. a comparison of outcomes between patients who go to inpatient rehabilitation and those who go directly home after surgery. Propensity based scoring and matching will be used to determine if outcomes are better in one of the two groups
2. determination of the predictors of the 'unhappy knee' 12 months post surgery. A case controlled matched design will be used.
3. comparison in satisfaction with the acute care experience between private and public patients in a subset
4. a comparison of outcomes between THR patients with an anterior surgical approach and a posterior approach
5. description of ambulation profiles immediately post surgery and variables associated with early ambulation
6. snapshot of rehabilitation received after TKA or THA

ELIGIBILITY:
Inclusion Criteria:

* Primary elective unilateral or bilateral total knee arthroplasty (TKA) or total hip arthroplasty (THA)
* Primary diagnosis of osteoarthritis
* Aged 18 or over, either gender
* Able to comprehend the protocol and provide consent (e.g. be able to read English, have no history of dementia)
* Available for telephone follow-up within the first 6 weeks, 3 months and then at 12 months post surgery
* No further joint replacement surgery planned within the next 3 months of the current surgery

Exclusion Criteria:

* Cognitive impairment / history of dementia
* Hip replacement for fracture
* Revision of previous joint replacement
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary total hip or knee replacement in private or public hsopitals in Australia
Sampling Method: Probability Sample
Enrollment: 1900 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Percentage of participants experiencing the composite outcome up to 35 days post surgery. | 35 days post total hip or knee replacement surgery
  The proportion of patients in each group (compliant and non-compliant groups) that experience one or more of the following outcomes - death, readmission, reoperation or surgical complication - up to 35 days post-surgery. Analyses will adjust for patient and service provider confounders.

SECONDARY OUTCOMES:
Patient-reported quality of life | 35 days post surgery
  The EuroQual 5-level (EQ5D) assessment will be used to capture patient-reported quality of life.
Incidence of venous thromboembolism | 90 days post surgery
  The number of patients treated with a documented blood clot
Incidence of deep infection. | 365 days post surgery
  The number of patients with a documented deep infection. That is, were treated with intravenous antibiotics for their index joint, was readmitted to hospital, and/or had a joint washout.
Costs of care processes | 90 days post surgery
  The cost of individual care processes, the cost of healthcare utilisation post discharge from acute care, carer costs and cost of time off work will be calculated for each person. Data will be collected using patient diaries and derived from the acute care study data.
Patient reported quality of life (QoL) | 90 days post surgery
  The EQ5D will be used to capture patient-reported QoL
Health-related QoL | 365 days post surgery
  The EQ5D will be used to capture QoL
Patient reported joint pain and function | 90 days post surgery
  The Oxford Knee or Hip Score will be used to capture patient reported joint specific pain and function.
Patient reported joint pain and function | 365 days post surgery
  The Oxford Knee or Hip Score will be used to capture patient reported joint specific pain and function

OTHER OUTCOMES:
Day of first ambulation attempt post surgery | day 0-14 post-surgery
  The first post-operative day the patient walked, including any partial or full weight-bearing activities such as walking on the spot, bed-to-chair and bed-to-toilet).
  first post-operative day that patients walked, including any partial or full weight-bearing activities 134
  such as walking on the spot, bed-to-chair and bed-to-toilet).

CONTACTS AND LOCATIONS:
Overall Officials: Justine M Naylor, PhD,BAppSc (Phty), Principal Investigator — Sydney South West Local health District, University of NSW, Ingham Institute for Applied Medical Research; Ian A Harris, PhD,MBBS, Principal Investigator — Sydney South West Local health District, University of NSW, Ingham Institute for Applied Medical Research; Helen M Badge, MApSc,BAScOT, Principal Investigator — Ingham Institute for Applied Medical Research, University of NSW; Wei Xuan, PhD, Principal Investigator — Ingham Institute Applied Medical Research; Christine Lin, PhD, BApScPhty, Principal Investigator — George Institute, University of Syndey, Australia; Elizabeth Armstrong, BAppScPhty, Principal Investigator — University of NSW, Sydney, Australia; Kevin Bozic, MD MBA, Principal Investigator — University of California, San Francisco; John Fletcher, PhD, MBBS, Principal Investigator — University of Sydney, Australia; Iain Gosbell, PhD, MBBS, Principal Investigator — University of Western Sydney, Australia
Locations (18):
- Australia (18):
  - Concealed site 4 Public, Rural, New South Wales
  - Concealed site 6 Private, Rural, New South Wales
  - Concealed site 8 Private, Rural, New South Wales
  - Concealed site 16 Public, Semi Rural, New South Wales
  - Concealed site 1 Public, Sydney, New South Wales
  - Concealed site 17 Private, Sydney, New South Wales
  - Concealed site 2 Public, Sydney, New South Wales
  - Concealed Site 3 Public, Sydney, New South Wales
  - Concealed site 5 Private, Sydney, New South Wales
  - Concealed site 7 Private, Urban, New South Wales
  - Concealed site 15 Public, Rural, Queensland
  - Concealed site 13 Private, Urban, Queensland
  - Concealed site 14 Public, Urban, Queensland
  - Concealed site 12 Private, Urban, South Australia
  - Concealed site 11 Private, Urban, Tasmania
  - Concealed site 9 Private, Melbourne, Victoria
  - Concealed site 10 Public, Urban, Victoria
  - Concealed site 18 - 2 Public sites, Urban, Victoria

REFERENCES:
- [Derived] Johns N, Naylor J, McKenzie D, Brady B, Olver J. High pain reported at 3 months post-total knee arthroplasty often persists for the next 3 years and is associated with reduced function and quality of life. Musculoskeletal Care. 2024 Mar;22(1):e1866. doi: 10.1002/msc.1866. PMID 38348944
- [Derived] Sidhu V, Badge H, Churches T, Maree Naylor J, Adie S, A Harris I. Comparative effectiveness of aspirin for symptomatic venous thromboembolism prophylaxis in patients undergoing total joint arthroplasty, a cohort study. BMC Musculoskelet Disord. 2023 Aug 3;24(1):629. doi: 10.1186/s12891-023-06750-x. PMID 37537580
- [Derived] Jenkin DE, Harris IA, Descallar J, Naylor JM. Discharge to inpatient rehabilitation following arthroplasty is a strong predictor of persistent opioid use 90 days after surgery: a prospective, observational study. BMC Musculoskelet Disord. 2023 Jan 14;24(1):31. doi: 10.1186/s12891-023-06142-1. PMID 36639624
- [Derived] Johns N, Naylor J, McKenzie D, Brady B, Olver J. Is inpatient rehabilitation a predictor of a lower incidence of persistent knee pain 3-months following total knee replacement? A retrospective, observational study. BMC Musculoskelet Disord. 2022 Sep 12;23(1):855. doi: 10.1186/s12891-022-05800-0. PMID 36096816
- [Derived] Naylor JM, Hart A, Mittal R, Harris IA, Xuan W. The effectiveness of inpatient rehabilitation after uncomplicated total hip arthroplasty: a propensity score matched cohort. BMC Musculoskelet Disord. 2018 Jul 18;19(1):236. doi: 10.1186/s12891-018-2134-3. PMID 30021552